CLINICAL TRIAL: NCT01830673
Title: Investigation of T-regulatory Cells After Subcutaneous Immunotherapy
Brief Title: Regulatory T-cells After Subcutaneous Immunotherapy
Acronym: RTCAS
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Dr. med. Martin Rosewich, Principal Investigator, Johann Wolfgang Goethe University Hospital
Other Study IDs: FRA-2012-SCIT
Record Dates: First submitted 2012-11-20; First posted 2013-04-12 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Grass Pollen Allergy; Specific Immunotherapy
Keywords: T-regulatory cells; TH1, TH2 cells; specific IgE; specific IgG; specific IgG4; IL2; IL5; IL10; IL12/23; Y-IFN; TNF-a

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- under SIT: patients completed second or third year of SIT. We include the patients directly after last SIT vaccination.
- after SIT: Patients completed three years of SIT for at least three years. We included them as a follow up.
- no SIT: These patients were determined randomly. They have a clinically relevant grass pollen allergy. They never had a SIT.

SUMMARY:
The primary endpoint was the induction of T-regulatory cells under s specific subcutaneous immunotherapy (SCIT). Patients suffering from grass pollen allergy (relevant clinical symptomes during the pollen season, Skin Prick test diamter >4mm or RAST class II or higher) were included. The patients were allocated to three study groups:

Group 1: during and directly after SCIT (after completion the 2nd or 3rd year of treatment) Group 2: completed SCIT more then three years ago Group 3: Patients with clinically relevant grass pollen allergy without SCIT.

The investigators analyzed the lung function parameters, exhaled NO (eNO) and asked the patients to record symptoms during the adjacent pollen season. A blood sample was drawn to analyze the amount of TH1 and TH2 and regulatory T-cells, inflammatory markers(IL-2, IL-5, IL-10, IL-12/23, TNF-alpha, IFN-gamma) and blocking antibodies (IgG, IgG4).

ELIGIBILITY:
Inclusion Criteria:

* informed consent,
* clinically relevant grass pollen allergy,
* age > 6 and < 28

Exclusion Criteria:

* severe unstable asthma,
* regular ingestion of antihistamine,
* systemic steroid therapy,
* lung funtcion VC < 70%,
* FEV1 < 65%

Ages: 7 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients aged 7-28 years of age with house grass pollen allergy
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2011-10; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Induction of regulatory t-cells | group 1: on average within one week after 4th injection of SCIT, group 2: more than three years (3-4 years) after SCIT completion, group 3: no specific time point because there was no intervention
  Determination of T-reulatory cells by FACS (staining for fox p3).

SECONDARY OUTCOMES:
TH1-cells by FACS | group 1: on average within one week after 4th injection of SCIT, group 2: more than three years (3-4 years) after SCIT completion, group 3: no specific time point because there was no intervention
  Staining for CD3, CD4, CD183
Th-2 cells by FACS | group 1: on average within one week after 4th injection of SCIT, group 2: more than three years (3-4 years) after SCIT completion, group 3: no specific time point because there was no intervention
  Staining for CD3, CD4, CD 194
Inflammatory cytokines | group 1: on average within one week after 4th injection of SCIT, group 2: more than three years (3-4 years) after SCIT completion, group 3: no specific time point because there was no intervention
  Cytokines (Il-2, Il-5, Il-10, Il-12/23, IFN-gamma, TNF-alpha) were determined by cytometric bead assay
Questionnaire | During the pollen season - for group 1: pollen season directly after completion of SCIT therapy, group 2: same pollen season as group 1, three years after completion of a 3 year SCIT, group 3: same pollen season as group 1 and 2
  questionnaire to assess the quality of life (QoL), the clinical symptoms and medication scores during the SCIT adjacent pollen season.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zielen, Prof., Study Director — Johann Wolfgang Goethe University Hospital
Locations (1):
- Johann Wolfgang Goethe-university, Frankfurt/M, Hesse, Germany

REFERENCES:
- [Background] Zielen S, Kardos P, Madonini E. Steroid-sparing effects with allergen-specific immunotherapy in children with asthma: a randomized controlled trial. J Allergy Clin Immunol. 2010 Nov;126(5):942-9. doi: 10.1016/j.jaci.2010.06.002. Epub 2010 Jul 10. PMID 20624650
- [Background] Martin M, Michalek SM, Katz J. Role of innate immune factors in the adjuvant activity of monophosphoryl lipid A. Infect Immun. 2003 May;71(5):2498-507. doi: 10.1128/IAI.71.5.2498-2507.2003. PMID 12704121
- [Background] Drachenberg KJ, Heinzkill M, Urban E, Woroniecki SR. Efficacy and tolerability of short-term specific immunotherapy with pollen allergoids adjuvanted by monophosphoryl lipid A (MPL) for children and adolescents. Allergol Immunopathol (Madr). 2003 Sep-Oct;31(5):270-7. doi: 10.1016/s0301-0546(03)79195-2. PMID 14572416
- [Background] Rosewich M, Schulze J, Eickmeier O, Telles T, Rose MA, Schubert R, Zielen S. Tolerance induction after specific immunotherapy with pollen allergoids adjuvanted by monophosphoryl lipid A in children. Clin Exp Immunol. 2010 Jun;160(3):403-10. doi: 10.1111/j.1365-2249.2010.04106.x. Epub 2010 Mar 16. PMID 20345983
- [Background] Rosewich M, Schulze J, Fischer von Weikersthal-Drachenberg KJ, Zielen S. Ultra-short course immunotherapy in children and adolescents during a 3-yrs post-marketing surveillance study. Pediatr Allergy Immunol. 2010 Feb;21(1 Pt 2):e185-9. doi: 10.1111/j.1399-3038.2009.00953.x. Epub 2009 Dec 8. PMID 20003062